CLINICAL TRIAL: NCT04643080
Title: Effects of a 12-week Dairy-based Probiotic Dietary Intervention on Cognitive Performance, Emotional Well-being, and Inflammation in Older Adults
Brief Title: Dairy Based Probiotic Intervention and Cognitive, Emotional, and Inflammatory Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Idaho (Other)
Collaborators: Kansas State University (Other)
Responsible Party: Principal Investigator, Annie Roe, Principal Investigator, University of Idaho
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 18-203
Record Dates: First submitted 2020-11-16; First posted 2020-11-24 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Cognitive Decline; Cognitive Change; Inflammation; Emotions
Keywords: Probiotics; Cognition; Emotional Wellbeing; Inflammation; Older Adults; Yogurt
MeSH Terms: conditions — Cognitive Dysfunction; Inflammation | interventions — Yogurt

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Subjects were asked to avoid consuming fermented foods for 12 weeks.
- Yogurt (Experimental): Subjects were asked to consume 6 oz. of yogurt daily for 12 weeks.
  Interventions: Other: Yogurt

INTERVENTIONS:
Other: Yogurt — 6 oz. of a commercially available yogurt were provided daily for 12 weeks
  Arms: Yogurt

SUMMARY:
The purpose of this study was to determine the effect of dairy-based probiotics on cognitive function, emotional wellbeing, and inflammation. Subjects were assigned to either consume 6 oz of yogurt/day or abstain from consuming yogurt and other probiotic-containing foods for 12 weeks. Subjects completed baseline testing and 12-week follow-up testing consisting of a laboratory blood draw to assess inflammatory biomarkers, and a computerized assessment to evaluate cognitive and emotional wellbeing measures.

ELIGIBILITY:
Inclusion Criteria:

* ability to participate in a 12-week study
* at least 50 years of age
* not currently taking a probiotic dietary supplement
* willing to refrain from consuming probiotic dietary supplements or fermented foods for 12-weeks
* willing to have blood drawn twice
* willing to consume yogurt daily for 12 weeks

Exclusion Criteria:

-

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2019-03-07 (Actual); Primary Completion 2019-07-15 (Actual); Study Completion 2019-07-15 (Actual)

PRIMARY OUTCOMES:
Change in Fluid Cognition Composite from Baseline to 12-weeks | Change from baseline fluid cognition composite score at 12-weeks
  Subjects completed a battery of computerized cognitive assessments at baseline and 12-weeks, using the NIHToolbox for Assessment of Neurological and Behavioral Function application. The fluid cognition composite score was derived from scores on the Flanker Inhibitory Control and Attention Test, Dimensional Change Card Sort Test, Picture Sequence Memory Test, Pattern Comparison Processing Speed Test, and List Sorting Working Memory test.
Change in Executive Function from Baseline to 12-weeks | Change from baseline executive function test scores at 12 weeks
  Subjects completed a battery of computerized cognitive assessments at baseline and 12-weeks, using the NIHToolbox for Assessment of Neurological and Behavioral Function application. Executive function was assessed by the Flanker Inhibitory Control and Attention Test and the Dimensional Change Card Sort Test.
Change in Attention from Baseline to 12-weeks | Change from baseline attention test scores at 12 weeks
  Subjects completed a battery of computerized cognitive assessments at baseline and 12-weeks, using the NIHToolbox for Assessment of Neurological and Behavioral Function application. Attention was assessed by the Flanker Inhibitory Control and Attention Test.
Change in Working Memory from Baseline to 12-weeks | Change from baseline working memory test scores at 12 weeks
  Subjects completed a battery of computerized cognitive assessments at baseline and 12-weeks, using the NIHToolbox for Assessment of Neurological and Behavioral Function application. Working Memory was assessed by the List Sorting Working Memory test.
Change in Processing Speed from Baseline to 12-weeks | Change from baseline processing speed test scores at 12 weeks
  Subjects completed a battery of computerized cognitive assessments at baseline and 12-weeks, using the NIHToolbox for Assessment of Neurological and Behavioral Function application. Processing Speed was assessed by the Pattern Comparison Processing Speed test.
Change in Episodic Memory from Baseline to 12-weeks | Change in baseline episodic memory score at 12 weeks
  Subjects completed a battery of computerized cognitive assessments at baseline and 12-weeks, using the NIHToolbox for Assessment of Neurological and Behavioral Function application. Episodic Memory was assessed by the Picture Sequence Memory test.

SECONDARY OUTCOMES:
Change in Negative Affect from Baseline to 12-weeks | Change from baseline negative affect test scores at 12 weeks
  Subjects completed a battery of computerized self-reported questionnaires using the NIHToolbox for Assessment of Neurological and Behavioral Function. A Negative Affect summary score was derived from 5 individual assessments of anger affect, anger hostility, sadness, fear affect, and perceived stress.
Change in Psychological Wellbeing | Change from baseline psychological satisfaction test scores at 12 weeks
  Subjects completed a battery of computerized self-reported questionnaires using the NIHToolbox for Assessment of Neurological and Behavioral Function. A Psychological Wellbeing summary score was derived from 3 individual assessments of life satisfaction, meaning, and positive affect.
Change in Social Satisfaction from Baseline to 12-weeks | Change from baseline social satisfaction test scores at 12 weeks
  Subjects completed a battery of computerized self-reported questionnaires using the NIHToolbox for Assessment of Neurological and Behavioral Function. A Social Satisfaction summary score was derived from 5 individual assessments of friendship, loneliness, emotional support, instrumental support, and perceived rejection.
Change in serum interleukin-6 concentration from baseline to 12 weeks | Change from baseline serum interleukin-6 concentration at 12 weeks
  Serum samples were analyzed to determine concentrations of interleukin-6 (pg/mL).
Change in serum tumor necrosis factor-alpha concentration from baseline to 12 weeks | Change from baseline serum tumor necrosis factor-alpha concentration at 12 weeks
  Serum samples were analyzed to determine concentrations of tumor necrosis factor-alpha (pg/mL).
Change in serum c-reactive protein concentration from baseline to 12 weeks | Change from baseline serum c-reactive protein concentration at 12 weeks
  Serum samples were analyzed to determine concentrations of c-reactive protein (mg/L).

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - University of Idaho, Boise, Idaho
  - University of Idaho, Coeur d'Alene, Idaho
  - University of Idaho, Pocatello, Idaho
  - Kansas State University, Manhattan, Kansas

IPD SHARING:
Plan to Share IPD: No
This is a small pilot study and there are not intentions to make individual participant data available to other researchers.